CLINICAL TRIAL: NCT06505161
Title: Dry Needling Versus Percutaneous Electrolysis in Lumbar Multifidus Muscles in Patients With Chronic Low Back Pain
Acronym: DN-PE-LBP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Leire López de Calle Sánchez, Leire López de Calle Sánchez, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dry needling Electrolysis
Record Dates: First submitted 2024-07-10; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Chronic Low-back Pain
Keywords: chronic low back pain; Dry needling; Percutaneous electrolysis
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: The subjects will be divided into two groups. The control group will receive DN treatment, and the experimental group will receive PE, both in the lumbar multifidus muscles.
Who Masked: Participant, Outcomes Assessor
Masking Description: 40 sealed opaque envelopes will be prepared. 20 of the envelopes will contain ballots corresponding to the DN control group and 20 to the PE group. Only the examiner who will carry out the intervention will know the group of each participant. The main examiner will be the one who monitors the intervention without knowing which group each participant belongs to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling group (Active Comparator): The dry needling group will recibe a dry needling treatment with the Hong technique.
  Interventions: Other: Dry needling
- Percutaneous electrolysis group (Experimental): The percutaneous electrolysis grupos will recibe a tratement of galvanic current at 1.5mA, with 3-5 impacts, for 3-5 seconds in the low back multifiud muscles.
  Interventions: Other: Percutaneous electrolysis

INTERVENTIONS:
Other: Dry needling — It consists in application of dry needling on active and/or latent TPs in low back multifidus muscles
  Arms: Dry needling group
Other: Percutaneous electrolysis — It consists in the application of intratissue percutaneous electrolysis with galvanic current as a cathodic flow electrode in the low back multifidus muscles. The intervention will be guided by ultrasound equipment medically certified.
  Arms: Percutaneous electrolysis group

SUMMARY:
The aim of this study is to evaluate the reduction of pain of two different treatments in patients with chronic low back pain. Patients were divided in two groups. The control group will receive DN treatment, and the experimental group will receive PE, both in the lumbar multifidus muscles.

DETAILED DESCRIPTION:
Background: Low back pain is one of the most common health problems and a leading cause of disability and absence from work. Between 70% and 80% of adults will experience an episode of low back pain and approximately 10.0% of them will become chronic. This has a direct impact on the lumbar stabilizing muscles, giving rise to both structural and functional changes. Among the different treatment options, it has been observed that both dry needling (DN) and percutaneous electrolysis (PE) are effective techniques in the management of musculoskeletal pain.

Aim: To evaluate whether the reduction of pain after the application of PE is superior to the one obtained with DN.

Methods: A single-blind randomized clinical trial will be conducted in patients with chronic low back pain. The subjects will be divided into two groups. The control group will receive DN treatment, and the experimental group will receive PE, both in the lumbar multifidus muscles. The study variables will be: pain (VAS), disability index (Oswestry Scale), fear of movement (TSK-11SV) and quality of life (SF-12). The measurements will be assessed before, right after and 7 days after a single intervention.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain ≥ 3 months.
* Age between 30 and 60 years old.
* Not being receiving other physical therapy

Exclusion Criteria:

* Diagnosis of specific lumbar pathology.
* History of previous lumbar surgery.
* Treatment with corticosteroids, anti-inflammatory or antibiotic medication in recent weeks.
* Oncological processes, febrile symptoms or thrombophlebitis.
* Skin conditions.
* Belonephobia.
* Pacemaker.
* Pregnancy.
* Patients with neurological pathology

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity. Visual analogue scale. | At baseline, at 1 week after the last intervention, and 6-month follow-up period
  A 10-point Numerical Pain Scale (0: no pain, 10: maximum pain) assesses the intensity of pain

SECONDARY OUTCOMES:
Disability. Oswestry Low Back Pain Disability Idex | At baseline, at 1 week after the last intervention, and 6-month follow-up period
  It has 10 items associated to activities of daily living, each item has a punctuation from 0 to 5 points
Fear of Movement. Tampa Scale of kinesiophobia (TSK-11SV) | At baseline, at 1 week after the last intervention, and 6-month follow-up period
  Is a 11-item questionnaire that measures the fear of movement and (re)injury.
Quality of life. SF-12 Health questionnaire. | At baseline, at 1 week after the last intervention, and 6-month follow-up period
  SF-12 Health questionnaire scores range from 0 to 100% and indicate the self-perceived health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Leire Lopez de Calle Sánchez, Grade, Principal Investigator — University of Alcala; Samuel Fernandez Carnero, PhD, Study Director — University of Alcala
Locations (1):
- Campus Científico-Tecnológico UAH. Av. de León, 3A, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ng SK, Urquhart DM, Fitzgerald PB, Cicuttini FM, Hussain SM, Fitzgibbon BM. The Relationship Between Structural and Functional Brain Changes and Altered Emotion and Cognition in Chronic Low Back Pain Brain Changes: A Systematic Review of MRI and fMRI Studies. Clin J Pain. 2018 Mar;34(3):237-261. doi: 10.1097/AJP.0000000000000534. PMID 28719509
- [Background] Chou R, Qaseem A, Snow V, Casey D, Cross JT Jr, Shekelle P, Owens DK; Clinical Efficacy Assessment Subcommittee of the American College of Physicians; American College of Physicians; American Pain Society Low Back Pain Guidelines Panel. Diagnosis and treatment of low back pain: a joint clinical practice guideline from the American College of Physicians and the American Pain Society. Ann Intern Med. 2007 Oct 2;147(7):478-91. doi: 10.7326/0003-4819-147-7-200710020-00006. PMID 17909209
- [Background] Matheve T, Hodges P, Danneels L. The Role of Back Muscle Dysfunctions in Chronic Low Back Pain: State-of-the-Art and Clinical Implications. J Clin Med. 2023 Aug 24;12(17):5510. doi: 10.3390/jcm12175510. PMID 37685576
- [Background] Hodges PW, Danneels L. Changes in Structure and Function of the Back Muscles in Low Back Pain: Different Time Points, Observations, and Mechanisms. J Orthop Sports Phys Ther. 2019 Jun;49(6):464-476. doi: 10.2519/jospt.2019.8827. PMID 31151377
- [Background] Hu HT, Gao H, Ma RJ, Zhao XF, Tian HF, Li L. Is dry needling effective for low back pain?: A systematic review and PRISMA-compliant meta-analysis. Medicine (Baltimore). 2018 Jun;97(26):e11225. doi: 10.1097/MD.0000000000011225. PMID 29952980
- [Background] Fakontis C, Iakovidis P, Lytras D, Kasimis K, Koutras G, Ntinou SR, Kottaras A, Chatziprodromidou IP, Chatzikonstantinou P, Apostolou T. Efficacy of percutaneous needle electrolysis versus dry needling in musculoskeletal pain: A systematic review and meta-analysis. J Back Musculoskelet Rehabil. 2023;36(5):1033-1046. doi: 10.3233/BMR-220408. PMID 37458028
- [Background] Valera-Calero JA, Sanchez-Mayoral-Martin A, Varol U. Short-term effectiveness of high- and low-intensity percutaneous electrolysis in patients with patellofemoral pain syndrome: A pilot study. World J Orthop. 2021 Oct 18;12(10):781-790. doi: 10.5312/wjo.v12.i10.781. eCollection 2021 Oct 18. PMID 34754834